CLINICAL TRIAL: NCT05908292
Title: Optimizing Postpartum Pelvic Health Through Self-Scar Tissue Massage of Episiotomy and Perineal Scar Tissue The EPIS Trial: A Pilot Randomized Control Trial to Determine Feasibility
Brief Title: Optimizing Postpartum Pelvic Health Through Self-Scar Tissue Massage of Episiotomy and Perineal Scar Tissue A Pilot RCT
Acronym: EPIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Alberta Health services (Other); Alberta Innovates Health Solutions (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: REB23-0097
Record Dates: First submitted 2023-05-15; First posted 2023-06-18 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-05

CONDITIONS: Episiotomy; Complications; Scar Tissue; Perineal Tear; Vaginal Tear Resulting From Childbirth
Keywords: Perineal Tear; Vaginal Tear; Episiotomy
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Episiotomy and Vaginal/Perineal Tear Self-Scar Massage (Experimental): This Arm will be instructed in and perform self-scar massage to their pelvic floor scar tissue.
  Interventions: Procedure: Pelvic Floor Scar Tissue Self-Scar Massage
- Standard Postnatal Care (No Intervention): This Arm will not be instructed in or perform self-scar massage to their pelvic floor scar tissue.

INTERVENTIONS:
Procedure: Pelvic Floor Scar Tissue Self-Scar Massage — Self scar-massage intervention of healed pelvic floor scar tissue for 5 minutes, 3x/week for 6 weeks.
  Arms: Episiotomy and Vaginal/Perineal Tear Self-Scar Massage

SUMMARY:
The goal of this Pilot Randomized Control Trial (RCT) is to determine if a larger RCT evaluating the effect of self-scar tissue massage of episiotomy and/or vagina/perineal tear scar tissue on pelvic health outcomes is feasible.

The main questions it aims to answer are:

Can the investigators recruit 130 participants and aim for 80% retention of participants in this study?

Are the response rates to questionnaires and completeness of questionnaires acceptable?

Do the participants find the self-scar tissue massage intervention easy and acceptable to perform and do they adhere to the protocol?

Type of Study: Clinical Trial

Participant Population/Health Conditions: The participant population will be 18 years of age or older, primiparous, within 1 year postpartum after vaginal delivery with healed episiotomy and/or vaginal perineal tear(s) as confirmed to them by their maternity care provider or family doctor at their 6 week postpartum check or other appointment. The participants will also need to have sufficient proficiency in English to understand intervention instructional video and complete written questionnaires.

Investigators will compare the scores on two reliable and validated pelvic health questionnaires in those in the intervention and control groups. The intervention group will be provided an instructional video on self-scar tissue massage and asked to perform self-scar massage and record their intervention and experience over a 6-week period. The control group will receive routine postnatal care (no self-scar massage training or performance). Patient medical records will be used to collect demographic data and labour and delivery characteristics. Two reliable and validated pelvic health questionnaires will be used for outcome measures. Baseline outcomes will be performed at the start of the study and then repeated 6 weeks later and again 18 weeks later.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Primiparous
* Within 1 year postpartum after vaginal delivery with episiotomy and/or vaginal/perineal tear
* Healed episiotomy and/or vagina/perineal tear as confirmed to them by their maternity care provider or family doctor at their postpartum check or other appointment
* Sufficient proficiency in English to understand intervention instructional video and complete written questionnaires.

Exclusion Criteria:

* Self-reported current vaginal infection or urinary tract infection
* Self-reported gynecological surgery after delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Rate of Participant Recruitment | 1 year
  To evaluate the rate of participant recruitment, the investigators will calculate how many participants were recruited on average per month per hospital site.
Rate of Participant Attrition | 1 year
  To evaluate the rate of participant attrition, the investigators will calculate the number of participants that drop out of the study over the total number of participants that are randomized in the study over the study period.
Number of Pelvic Floor Distress Inventory (PFDI-20) Outcome Measures with missing data | 1 year
  To evaluate the response rate and the completeness of the PFDI-20 the investigators will track how many questionnaires are not completed and determine if there is any missing data in the responses to the PFDI-20.
Number of The Carol Scale with missing data | 1 year
  To evaluate the response rate and the completeness of the Carol Scale the investigators will track how many questionnaires are not completed and determine if there is any missing data in the responses to the Carol Scale.
Number of participants to complete self-scar massage protocol as intended | 1 year
  To evaluate the acceptability of the self-scar massage intervention, the investigators will examine participants' reported intervention frequency and time of intervention on their records and note any deviation from the intervention protocol. Some participant interviews will be conducted from a program evaluation lens to determine how the intervention was received. Exemplar quotes will be used to describe participants experience of the self-scar massage intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Brennand, MD, MSc, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No